CLINICAL TRIAL: NCT03065023
Title: A Phase I/II, Multicenter, Open-label, Clinical Trial of Intratumoral/Intralesional Administration of RGT100 in Subjects With Advanced or Recurrent Tumors
Brief Title: Study of Intralesional Administration of MK-4621 (RGT100) in Adult Participants With Advanced or Recurrent Tumors (MK-4621-001/RGT100-001)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Group B not started for business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4621-001; 2016-003028-22 (EudraCT Number); RGT100-001 (Other: Rigontec GMBH); MK-4621-001 (Other: Merck)
Record Dates: First submitted 2017-02-10; First posted 2017-02-27 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced tumor; Intratumoral injection; Intralesional injection

STUDY DESIGN:
Intervention Model Description: The study was to be conducted in 2 groups:
  * Group A: participants with transdermally/transmucosally injectable tumors, and
  * Group B: participants with injectable liver tumors or liver metastases. However, Group B was not started.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Cutaenous lesions (Experimental): Participants with transdermally/transmucosally injectable tumors including cutaneous, subcutaneous or lymph node injectable tumors received escalating doses of MK-4621 via intratumoral (IT)/intralesional (IL) injection twice each week (Q2W) over a period of 4 weeks. Participants may have continued to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (up to approximately 2 years).
  Interventions: Drug: MK-4621
- Group B: Liver lesions (Experimental): Participants with injectable liver tumors or liver metastases were to receive escalating doses of MK-4621 via intratumoral (IT)/intralesional (IL) injection once each week over a period of 4 weeks. Participants were to have been able to continue to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (up to approximately 2 years). (Group B was not started. Development will continue with new protocol.)
  Interventions: Drug: MK-4621

INTERVENTIONS:
Drug: MK-4621 — IT/IL injection Fixed concentration of 0.2 mg/mL Starting dose: 0.2 mg
  Other Names: RGT100

SUMMARY:
This is a Phase I/II multicenter, first-in-human open-label, dose escalation study to evaluate the safety, tolerability, and anti-tumor activity of intratumoral (IT)/intralesional (IL) injections of MK-4621 (RGT100) in adult participants with selected advanced or recurrent tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years
2. Participants with histologically or cytologically confirmed diagnosis of advanced or recurrent tumors (including lymphomas) for whom all standard treatments have been used or are not feasible and MK-4621 (RGT100) is a suitable treatment option and:

   1. For Group A: has cutaneous, sub-cutaneous (SC), or lymph node injectable tumors
   2. For Group B: has injectable liver tumors or liver metastases
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Life expectancy >3 months as assessed by the Investigator
5. Adequate organ function
6. Negative serum pregnancy test within 2 weeks before first dose of study drug if the participant is a woman of childbearing potential. Participants and participant's partners of childbearing potential must agree to use birth control consistently and correctly during the study and for at least 6 months after the last study drug application.
7. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and 1 separate injectable lesion with diameter ≥1 cm but <7 cm
8. Ability to provide written informed consent before any study drug-related screening procedures being performed

Exclusion Criteria:

1. Any tumor-directed therapy within 4 weeks before study treatment
2. Treatment with investigational drugs within 4 weeks before study enrolment
3. Systemic steroids at a dose of >10 mg of prednisolone, >2 mg of dexamethasone a day or equivalent, except topical (inhaled, topical, nasal) for the last 28 days and ongoing
4. Participants with rapidly progressing disease (as determined by the Investigator)
5. Ongoing immune-related adverse events (irAEs) and/or adverse events (AEs) ≥ grade 2 not resolved from previous therapies except vitiligo, stable neuropathy grade 2, hair loss, and stable endocrinopathies with substitutive hormone therapy
6. Within 4 weeks of major surgery
7. Prior splenectomy
8. Documented history of active autoimmune disorders requiring systemic immunosuppressive therapy
9. Primary or secondary immune deficiency
10. Active allergy requiring systemic medication or active infections requiring anti-infectious therapy
11. Seropositive (except after vaccination) for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
12. Clinically significant cardiac disease including heart failure (New York Heart Association, Class III or IV), pre-existing arrhythmia, uncontrolled angina pectoris, or myocardial infarction within 1 year before study entry
13. Dementia or altered mental status that would prohibit informed consent
14. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study assessed by the Investigator
15. History of stroke, seizures, encephalitis, or multiple sclerosis
16. Gastric ulcer or inflammatory bowel disease or Crohn's disease or ulcerative colitis in the last 6 months
17. Active drug or alcohol abuse
18. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus - Phase I Unit, Dresden
  - Universitätsklinikum Essen, Essen
  - National Center for Tumor Diseases, Heidelberg
- Spain (2):
  - START - Fundación Jiménez Díaz - Phase I Unit, Madrid
  - START - Hospital Universitario HM Sanchinarro - Phase I Unit, Madrid
- University of Oxford Department of Oncology, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Moreno V, Calvo E, Middleton MR, Barlesi F, Gaudy-Marqueste C, Italiano A, Romano E, Marabelle A, Chartash E, Dobrenkov K, Zhou H, Connors EC, Zhang Y, Wermke M. Treatment with a retinoic acid-inducible gene I (RIG-I) agonist as monotherapy and in combination with pembrolizumab in patients with advanced solid tumors: results from two phase 1 studies. Cancer Immunol Immunother. 2022 Dec;71(12):2985-2998. doi: 10.1007/s00262-022-03191-8. Epub 2022 May 21. PMID 35596791

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: MK-4621 0.2 mg: Participants with transdermally/transmucosally injectable tumors including cutaneous, subcutaneous or lymph node injectable tumors received MK-4621 0.2.mg via intratumoral (IT)/intralesional (IL) injection twice each week over a period of 4 weeks during Cycle 1. Participants may have continued to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (could have been up to approximately 2 years). Each cycle was 28 days.
- Group A: MK-4621 0.4 mg: Participants with transdermally/transmucosally injectable tumors including cutaneous, subcutaneous or lymph node injectable tumors received MK-4621 0.4 mg via IT/IL injection twice each week over a period of 4 weeks during Cycle 1. Participants may have continued to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (could have been up to approximately 2 years). Each cycle was 28 days.
- Group A: MK-4621 0.6 mg: Participants with transdermally/transmucosally injectable tumors including cutaneous, subcutaneous or lymph node injectable tumors received MK-4621 0.6 mg via IT/IL injection twice each week over a period of 4 weeks during Cycle 1. Participants may have continued to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (could have been up to approximately 2 years). Each cycle was 28 days.
- Group A: MK-4621 0.8 mg: Participants with transdermally/transmucosally injectable tumors including cutaneous, subcutaneous or lymph node injectable tumors received MK-4621 0.8 mg via IT/IL injection twice each week over a period of 4 weeks during Cycle 1. Participants may have continued to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (could have been up to approximately 2 years). Each cycle was 28 days.
- Group B: Liver Lesions: Participants with injectable liver tumors or liver metastases were to receive escalating doses of MK-4621 via IT/IL injection once each week over a period of 4 weeks. Participants were to have been able to continue to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (could have been up to approximately 2 years). (Group B was not started for business reasons. Development will continue with new protocol.)
Period: Overall Study
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg | Group B: Liver Lesions
Started | 3 | 3 | 3 | 6 | 0 (Group B not started for business reasons.)
Completed | 1 | 1 | 2 | 3 | 0
Not Completed | 2 | 2 | 1 | 3 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Participant Decision | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: MK-4621 0.2 mg: Participants with transdermally/transmucosally injectable tumors including cutaneous, subcutaneous or lymph node injectable tumors received MK-4621 0.2.mg via IT/IL injection twice each week over a period of 4 weeks during Cycle 1. Participants may have continued to receive study treatment beyond Cycle 1 for the remaining duration of the study as long as clinical benefit (no overt clinical progression or toxicity considered to be intolerable as per Investigator's assessment) was present (could have been up to approximately 2 years). Each cycle was 28 days.
- Total: Total of all reporting groups
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (26.8) | 48.7 (18.1) | 55.3 (16.0) | 64.2 (8.3) | 56.8 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 7
  Male | 1 | 2 | 1 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 6 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Plasma Cytokine Release by Cytokine Type [Median (Full Range); unit: ng/L] — Blood samples were collected at baseline for the analysis of cytokine release for selected cytokines (Interleukin-6 [IL-6] & tumor necrosis factor-alpha [TNF-a]) in plasma. (IL-6 Lower Limit of Quantification [LLOQ]: 9.3 ng/L & 7.5 ng/L for the 2 lower doses & the 2 higher doses, respectively. TNF-a LLOQ: 8.3 ng/L & 9.7 ng/L for the 2 lower doses & for the 2 higher doses, respectively.)
  ng/L
    IL-6 | 9.3 [9.3 to 9.3] | 9.3 [9.3 to 31.5] | 10 [7.5 to 12.9] | 7.5 [7.5 to 15.6] | 9.3 [7.5 to 31.5]
    TNF-a | 8.3 [8.3 to 8.3] | 8.3 [8.3 to 8.3] | 24.2 [9.7 to 24.4] | 9.7 [9.7 to 30.4] | 9.7 [8.3 to 30.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-related Adverse Event (AE) or Laboratory Abnormality by Severity Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 Criteria
Description: An AE was defined as any untoward medical occurrence in a study participant administered study treatment which did not necessarily have a causal relationship with this treatment. Treatment-related was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator. Severity of AE referred to the extent to which an AE affected the participants daily activities as assessed by the Investigator and was based on NCI CTCAE grades: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe or medically significant but not immediately life-threatening); Grade 4 (Life-threatening consequences); or Grade 5 (Death related to AE). The number of participants who experienced at least one treatment-related AE or laboratory abnormality are presented by severity.
Time Frame: Up to 90 days post last injection (Up to approximately 192 days)
Population: The safety population consisted of all participants who received ≥1 injection of MK-4621.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants
  Grade 1 | 1 | 2 | 2 | 3
  Grade 2 | 0 | 1 | 1 | 2
  Grade 3 | 1 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Description: A SAE was defined as any AE, regardless of dose, causality or expectedness, that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolonged existing inpatient hospitalization;
  * Resulted in persistent or significant incapacity or disability;
  * Was a congenital anomaly or birth defect; or
  * Was any other medically important event.
Time Frame: Up to 90 days post last injection (Up to approximately 192 days)
Population: The safety population consisted of all participants who received ≥1 injection of MK-4621.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 2 | 2 | 1 | 3

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to a Treatment-related Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a study participant administered a study treatment which did not necessarily have a causal relationship with this treatment. Treatment-related was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator. The number of participants who discontinued study treatment due to a treatment-related AE is presented.
Time Frame: Up to last injection (Up to approximately 102 days)
Population: The safety population consisted of all participants who received ≥1 injection of MK-4621.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT) by Severity Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 Criteria
Description: DLTs were assessed during the first treatment cycle (28 days) & were defined as any drug-related toxicity that occurred during the 28-day DLT period and included:
  * Non-hematologic toxicity grade ≥3 (except diarrhea, nausea, and vomiting unless lasting >3 days despite optimal supportive care);
  * Confirmed (with a second measurement after 24 hours) non-hematologic appropriately graded laboratory findings of Grade ≥3 that were ≤ Grade 1 at baseline;
  * Hematologic toxicity:
    * Grade 4 neutropenia ≥5 days, or Grade 3 neutropenia with fever (fever is >38.4ºC)
    * Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia lasting >7 days or with bleeding; and
  * Any other toxicity assessed as related to MK-4621, and which, in the opinion of the Investigator and the Sponsor physician constituted a DLT.
  The number of participants who experienced a DLT is presented by NCI CTCAE version 4.03 severity grade.
Time Frame: Cycle 1 (Up to approximately 28 days); Each cycle was 28 days.
Population: The DLT evaluable population consisted of participants who completed Cycle 1 (Day 28) or withdrew early for experiencing a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

5. Secondary Outcome: Objective Response Rate as Evaluated Radiologically Using Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR) or a Partial Response. Per irRECIST, CR (irCR) was defined as the complete disappearance of all measurable and non-measurable lesions. Lymph nodes must also have decreased to <0 mm in short axis. And, per irRECIST, Partial Response (irPR) was defined as a decrease of ≥30% in total measured tumor burden (TMTB) relative to baseline. For this study, irRECIST was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced an irCR or irPR based on irRECIST is presented.
Time Frame: Up to 60 days post last injection (Up to approximately 162 days)
Population: The efficacy population consisted of all allocated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Percentage of Participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 45.9]

6. Other Pre Specified Outcome: Mean Fold Change From Baseline in Plasma Cytokine Release by Cytokine Type: Day 1 (6 Hours Post Injection)
Description: Blood samples were collected at various time points for the analysis of mean fold change from baseline in cytokine release for selected cytokines (Interleukin-6 [IL-6] and tumor necrosis factor-alpha [TNF-a]) in plasma.
Time Frame: Baseline and Cycle 1 Day 1 (6 hours post injection) (Up to 1 day); Each cycle was 28 days.
Population: The cytokine evaluable population consisted of all participants who received ≥1 dose of MK-4621 and had baseline and post treatment cytokine data.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Fold change
  IL-6 | 1 (0) | 1.95 (1.64) | 2.71 (2.34) | 2.52 (3.14)
  TNF-a | 1 (0) | 1 (0) | 1 (0.6) | 0.89 (0.28)

7. Other Pre Specified Outcome: Mean Fold Change From Baseline in Plasma Cytokine Release by Cytokine Type: Day 1 (24 Hours Post Injection)
Description: as for outcome 6
Time Frame: Baseline and Cycle 1 Day 1 (24 hours post injection) (Up to 2 days); Each cycle was 28 days.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 2 | 3 | 3 | 6
Fold change
  IL-6 | 1 (0) | 1.27 (0.46) | 1.14 (0.3) | 1.68 (0.97)
  TNF-a | 1 (0) | 1 (0) | 1.48 (1.44) | 0.89 (0.28)

8. Other Pre Specified Outcome: Mean Fold Change From Baseline in Plasma Cytokine Release by Cytokine Type: Day 25 (6 Hours Post Injection)
Description: as for outcome 6
Time Frame: Baseline and Cycle 1 Day 25 (6 hours post injection) (Up to 25 days); Each cycle was 28 days.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 5
Fold change
  IL-6 | 0.95 (0.08) | 2 (1.11) | 1.02 (0.31) | 1.5 (0.61)
  TNF-a | 1 (0) | 1 (0) | 0.77 (0.21) | 0.77 (0.29)

9. Other Pre Specified Outcome: Mean Fold Change From Baseline in Plasma Cytokine Release by Cytokine Type: Day 25 (24 Hours Post Injection)
Description: as for outcome 6
Time Frame: Baseline and Cycle 1 Day 25 (24 hours post injection) (Up to 26 days); Each cycle was 28 days.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 5
Fold change
  IL-6 | 1.52 (0.9) | 1 (0) | 0.99 (0.1) | 0.89 (0.19)
  TNF-a | 1 (0) | 1 (0) | 1.02 (0.63) | 0.88 (0.32)

10. Other Pre Specified Outcome: Area Under the Concentration-Time Curve From Start of Dosing to Last Observed Concentration Above Limit of Quantitation (AUC0-t) of MK-4621: Day 1
Description: Blood samples were collected at various time points during Cycle 1 for the determination of MK-4621 AUC0-t on Day 1, which was defined as the AUC from the start time of dosing to the time of the last observed concentration above the limit of quantitation (LOQ).
Time Frame: Cycle 1 Day 1: Predose, 5 and 30 minutes, 2, 4, 6 and 24 hours post dose (Up to 2 days); Each cycle was 28 days.
Population: The pharmacokinetic evaluable population consisted of all participants who received ≥1 injection of MK-4621 and had pre- and post-treatment pharmacokinetic data for AUC0-t on Cycle 1 Day 1.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
h*ng/mL | 0.00 (0.00) | 0.174 (0.157) | 0.0360 (0.0623) | 1.87 (4.55)

11. Other Pre Specified Outcome: Area Under the Concentration-Time Curve From Start of Dosing to Last Observed Concentration Above Limit of Quantitation (AUC0-t) of MK-4621: Day 25
Description: Blood samples were collected at various time points during Cycle 1 for the determination of MK-4621 AUC0-t on Day 25, which was defined as the AUC from the start time of dosing to the time of the last observed concentration above the limit of quantitation (LOQ).
Time Frame: Cycle 1 Day 25: Predose, 5 and 30 minutes, 2, 4, 6 and 24 hours post dose (Up to 26 days); Each cycle was 28 days.
Population: The pharmacokinetic evaluable population consisted of all participants who received ≥1 injection of MK-4621 and had pre- and post-treatment pharmacokinetic data for AUC0-t on Cycle 1 Day 25.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 5
h*ng/mL | 0.00 (0.00) | 1.07 (0.767) | 0.099 (0.172) | 0.156 (0.350)

12. Other Pre Specified Outcome: Maximum Plasma Concentration (Cmax) of MK-4621: Day 1
Description: Blood samples were collected at various time points during Cycle 1 for the determination of MK-4621 Cmax on Day 1.
Time Frame: Cycle 1 Day 1: Predose, 5 and 30 minutes, 2, 4, 6 and 24 hours post dose (Up to 2 days); Each cycle was 28 days.
Population: The pharmacokinetic evaluable population consisted of all participants who received ≥1 injection of MK-4621 and had pre- and post-treatment pharmacokinetic data for Cmax on Cycle 1 Day 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
ng/mL | 0.00 (0.00) | 4.18 (3.76) | 0.863 (1.50) | 9.24 (21.9)

13. Other Pre Specified Outcome: Maximum Plasma Concentration (Cmax) of MK-4621: Day 25
Description: Blood samples were collected at various time points during Cycle 1 for the determination of MK-4621 Cmax on Day 25.
Time Frame: Cycle 1 Day 25: Predose, 5 and 30 minutes, 2, 4, 6 and 24 hours post dose (Up to 26 days); Each cycle was 28 days.
Population: The pharmacokinetic evaluable population consisted of all participants who received ≥1 injection of MK-4621 and had pre- and post-treatment pharmacokinetic data for Cmax on Cycle 1 Day 25.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 3 | 3 | 3 | 5
ng/mL | 0.00 (0.00) | 7.43 (2.44) | 1.703 (2.95) | 3.75 (8.39)

14. Other Pre Specified Outcome: Immune Infiltration of Injected Tumors by CD3 T Cell Receptor and Ki-67 Nuclear Protein: Day 1
Description: Sequential participant tumor biopsies were assessed via immunohistochemistry for the presence of tumor infiltrating CD3 T cell co-receptor-marked cells and Ki-67 nuclear protein-marked cells in tumor biopsies. CD3 is a marker of T cells and KI-67 is a cell marker of proliferation and activation. The percentage of positive CD3-marked cells and double-positive CD3 and Ki-67 nuclear protein-marked cells in tumor biopsies predose on Day 1 are presented.
Time Frame: Day 1 prior to injection (Up to 1 day)
Population: The immune infiltration evaluable population consisted of all participants who received ≥1 dose of MK-4621 and had pre- and post-treatment immune infiltration data.
Measure: Median (Full Range); unit: Percentage Positive Cells
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 1 | 3 | 1 | 1
Percentage Positive Cells
  CD3 Cells | 8.81 [8.81 to 8.81] | 17.58 [7.03 to 20.81] | 34.64 [34.64 to 34.64] | 17.34 [17.34 to 17.34]
  Ki-67 Positive CD3 Cells | 25.44 [25.44 to 25.44] | 25.19 [18.46 to 48.86] | 39.23 [39.23 to 39.23] | 32.19 [32.19 to 32.19]

15. Other Pre Specified Outcome: Immune Infiltration of Injected Tumors by CD3 T Cell Receptor and Ki-67 Nuclear Protein: Day 25
Description: Sequential participant tumor biopsies were assessed via immunohistochemistry for the presence of tumor infiltrating CD3 T cell co-receptor-marked cells and Ki-67 nuclear protein-marked cells in tumor biopsies. CD3 is a marker of T cells and KI-67 is a cell marker of proliferation and activation. The percentage of positive CD3-marked cells and double-positive CD3 and Ki-67 nuclear protein-marked cells in tumor biopsies postdose on Day 25 are presented.
Time Frame: Day 25 post injection (Up to 25 days)
Population: as for outcome 14
Measure: Median (Full Range); unit: Percentage Positive Cells
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
Number analyzed (Participants) | 1 | 3 | 1 | 1
Percentage Positive Cells
  CD3 Cells | 12.72 [12.72 to 12.72] | 8.43 [8.09 to 12.00] | 11.77 [11.77 to 11.77] | 32.19 [32.19 to 32.19]
  Ki-67 Positive CD3 Cells | 16.96 [16.96 to 16.96] | 36.39 [35.81 to 48.32] | 17.93 [17.93 to 17.93] | 12.16 [12.16 to 12.16]

ADVERSE EVENTS:
Time Frame: From first dose through up to 90 days after last dose (Up to approximately 192 days)
Description: Safety Population: All participants who received ≥1 injection of MK-4621. Per protocol, disease progression of cancer under study was not considered an adverse event (AE) unless considered related to study treatment. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Group A: MK-4621 0.2 mg | Group A: MK-4621 0.4 mg | Group A: MK-4621 0.6 mg | Group A: MK-4621 0.8 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 1/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: MK-4621 0.2 mg (N=3) | Group A: MK-4621 0.4 mg (N=3) | Group A: MK-4621 0.6 mg (N=3) | Group A: MK-4621 0.8 mg (N=6)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: MK-4621 0.2 mg (N=3) | Group A: MK-4621 0.4 mg (N=3) | Group A: MK-4621 0.6 mg (N=3) | Group A: MK-4621 0.8 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (6)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 3 (4) | 5 (8)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Group B not started for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the Investigator(s). Published data must not compromise the objectives of the study. Data from individual study sites in multicenter studies must not be published separately.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT03065023/Prot_SAP_000.pdf